CLINICAL TRIAL: NCT01675908
Title: Multicenter Randomized Trial Comparing Covered Metal and Plastic Stents for Preoperative Biliary Decompression in Pancreatic Cancer
Brief Title: Trial Comparing Metal Versus Plastic Stents for Preoperative Biliary Decompression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth (Other)
Collaborators: Vanderbilt University (Other); University of Maryland, Baltimore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 356090
Record Dates: First submitted 2012-08-28; First posted 2012-08-30 (Estimated); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Obstructive Jaundice; Pancreatic Cancer
MeSH Terms: conditions — Jaundice, Obstructive; Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metal stent (Active Comparator): Patients randomized to one cohort will undergo placement of fully covered self expandable metal stents. The rates (%) of stent dysfunction and complications will be evaluated.
  Interventions: Procedure: Stent Dysfunction; Procedure: Complications
- Plastic Stent (Active Comparator): At ERCP, a 10Fr plastic stent will be placed in the bile duct. The rates (%) of stent dysfunction and complications will be evaluated.
  Interventions: Procedure: Stent Dysfunction; Procedure: Complications

INTERVENTIONS:
Procedure: Stent Dysfunction — Rate of stent dysfunction (%) which includes persistent hyperbilirubinemia or cholangitis that warrant stent exchange by another ERCP.
Procedure: Complications — Rates of procedural complications (%) such as pancreatitis, perforation or hemorrhage during stent placement will be assessed.

SUMMARY:
Compare the performance of full covered metal stents and plastic stents for preoperative biliary decompression

DETAILED DESCRIPTION:
Covered self expandable metal stents (CSEMS) are three times larger in diameter than 10 Fr plastic stents. When compared to plastic stents, randomized trials have shown longer patency and fewer stent-related complications for CSEMS. The investigators hypothesize that placement of CSEMS would be a better treatment option for preoperative biliary decompression in patients with pancreatic cancer.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Patients with pancreatic cancer and mass in the head of pancreas causing jaundice.
2. Patients 19 yrs of age and older
3. Serum bilirubin > 2mg/dl
4. CT: No evidence of distant metastasis or local vascular invasion (tumor surrounding portal or mesenteric vessels for more than 180 degrees of their circumference or an irregular vessel margin).

EXCLUSION CRITERIA:

1. Karnofsky score < 60
2. Prior (ERCP or PTC) attempts at biliary decompression for the same indication
3. Tumor-related gastric outlet obstruction (vomiting and oral intake of < 1L/day)
4. Ongoing or planned neoadjuvant therapy
5. Cholangitis at presentation or coagulopathy needing reversal medication
6. Post-surgical anatomy
7. Multiple extra-hepatic biliary strictures or concomitant stricture in liver hilum
8. Failed ERCP's (Definition: Inability to deploy a biliary stent thereby requiring a PTC or surgery).

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2012-08-22 (Actual); Primary Completion 2019-08-21 (Actual); Study Completion 2019-08-21 (Actual)

PRIMARY OUTCOMES:
Complications related to stent dysfunction | 30 days
  Evaluate the rates of complications (%) related to stent dysfunction which include persistent hyperbilirubinemia and cholangitis that warrant stent exchange by a repeat ERCP.

SECONDARY OUTCOMES:
Procedural complications | 30 days
  This will be measured as proportion of patients who encounter a procedural complication (%) during ERCP that includes pancreatitis, perforation or hemorrhage.

CONTACTS AND LOCATIONS:
Overall Officials: shyam varadarajulu, MD, Principal Investigator — Florida Hospital Center for Interventional Endoscopy
Locations (1):
- Florida Hospital, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No
A manuscript will be developed following completion of the study.